CLINICAL TRIAL: NCT00948532
Title: Osteocel® Plus in eXtreme Lateral Interbody Fusion (XLIF®): Evaluation of Radiographic and Patient Outcomes
Brief Title: Osteocel® Plus in eXtreme Lateral Interbody Fusion (XLIF®)
Status: Completed | Type: Observational
Sponsor: NuVasive (Industry)
Responsible Party: Sponsor
Organization: Globus Medical Inc (Industry)
Other Study IDs: NUVA.OC.0801
Record Dates: First submitted 2009-07-16; First posted 2009-07-29 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Degenerative Disc Disease; Back Pain
Keywords: degenerative disc disease; lumbar spine; XLIF; Degenerative conditions
MeSH Terms: conditions — Intervertebral Disc Degeneration; Back Pain | interventions — Biological Products

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: biologic, Osteocel Plus — Osteocel® Plus
  Other Names: Osteocel® Plus

SUMMARY:
This is a prospective, non-randomized multi-center study to compare the use of Osteocel® Plus in subjects who receive XLIF® (eXtreme Lateral Interbody Fusion) surgery at one or two levels. These subjects will present with degenerative conditions in the lumbar spine that are amenable to surgical treatment and will be screened prior to study enrollment. Subjects will receive Osteocel Plus during their XLIF operation. Subjects will be followed for 24-months following surgery to determine the number of study subjects that are solidly fused at or before 24 months postoperatively, and to determine the mean time to fusion. This data will be compared to published and/or retrospective data for autograft, synthetic ceramics and Bone Morphogenetic Protein (BMP).

DETAILED DESCRIPTION:
Osteocel Plus is an allograft cellular bone matrix containing native mesenchymal stem cells (MSCs) which is intended to mimic the biologic performance of autograft without the morbidity associated with the autograft harvest. Mesenchymal stem cells, like those found in Osteocel Plus, are naturally occurring in the body and can differentiate into a variety of tissue types, depending on the local environment. Once implanted, MSCs can differentiate into osteoblasts, which produce new bone matrix. MSCs also naturally secrete bone-inducing growth factors that signal the patient's endogenous cells to migrate and participate in the bone formation process. Osteocel Plus is different from other orthobiologic products such as DBM and allograft cancellous bone because it contains living stem cells, which provide osteogenic potential. The cells include mesenchymal stem cells from an adult human donor; they are not from an embryonic source.

This study is being conducted to determine the percentage of patients with solid spinal fusions after being treated with Osteocel in an XLIF procedure. Due to the unique processing conditions, Osteocel Plus retains a high concentration of stem cells in conjunction with the allograft bone matrix, so it is hypothesized that the fusion rate with Osteocel Plus will be comparable to published data for autograft. The Osteocel product family has already been used in approximately 15,000 cases worldwide.

ELIGIBILITY:
Inclusion Criteria:

1. Persistent back and/or leg pain unresponsive to conservative treatment for at least six (6) months, unless clinically indicated earlier
2. Indicated for interbody fusion of one or two contiguous lumbar segments (L1 to L5)
3. Objective evidence of primary diagnosis must be confirmed by appropriate imaging studies
4. 18-80 years of age at the date of written informed consent
5. Able to undergo surgery based on physical exam, medical history and surgeon judgment
6. Expected to survive at least 2 years beyond surgery
7. Willing and able to return for post-treatment exams according to the follow-up called for in the protocol
8. Signed and dated Informed Consent Form

Exclusion Criteria:

1. Patient has a mental or physical condition that would limit the ability to comply with study requirements
2. Lumbar spine abnormality requiring treatment at more than two levels
3. Systemic or local infection; active or latent
4. Previous failed fusion at the operative level
5. Diseases that significantly inhibit bone healing (osteoporosis, metabolic bone disease, uncontrolled diabetes, dialysis dependent renal failure, symptomatic liver disease)
6. Undergoing chemotherapy or radiation treatment, or chronic use of steroids (defined as more than 6 weeks of steroid use within 12 months of surgery, other than episodic use or inhaled corticosteroids)
7. Pregnant, or plans to become pregnant during the study
8. Subject is a prisoner
9. Involvement in active litigation relating to the spine (worker's compensation claim is allowed if it is not contended)
10. A significant general illness (e.g., HIV, active metastatic cancer of any type) is present; subject is immunocompromised or is being treated with immunosuppressive agents
11. Participating in another clinical study that would confound study data

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Existing clinic patients
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2009-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects with radiographically apparent fusion. | 6-months, 12-months and 24-months

SECONDARY OUTCOMES:
The evaluation of angular displacement on flexion/extension films. | Post-op, 6-week, 3-month, 6-month, 12-month, 24-month
The evaluation of bridging bone on CT. | 6-month, 12-month
Preservation of interbody height over time. | All post-operative follow-up visits: Post-op, 6-week, 3-month, 6-month, 12-month, 24-month
The rate of complications attributable to the use of Osteocel Plus requiring intervention. | All study follow-up visits: Post-op, 6-week, 3-month, 6-month, 12-month, 24-month
The change in subject self-reported pain ratings (VAS scores). | from baseline through post-operation follow-up (visits at post-op, 6-week, 3-month, 6-month, 12-month and 24-months)
The change in Oswestry Disability Index scores. | from baseline through post-operation follow-up (visits at post-op, 6-week, 3-month, 6-month, 12-month and 24-months)

CONTACTS AND LOCATIONS:
Overall Officials: Kelli Howell, MS, Study Director — NuVasive
Locations (13):
- United States (13):
  - Shiley Center for Orthopaedic, Scripps Green Hospital, La Jolla, California
  - Broward Spine Institute, Hollywood, Florida
  - South Florida Spine Institute, Mount Sinai Medical Center, Miami Beach, Florida
  - Southeastern Spine Center, Doctors Hospital of Sarasota, Sarasota, Florida
  - USF, Tampa General Hospital, Tampa, Florida
  - Pinnacle Orthopaedics, Wellstone Kennestone Hospital, Marietta, Georgia
  - The Spine Center of DuPage Medical Group, Edward Hospital, Naperville, Illinois
  - Indiana Center for Neurosurgery, Indianapolis, Indiana
  - Columbia Orthopaedic Group, Boone Hospital Center, Columbia, Missouri
  - Spine Midwest, St. Mary's Health Center, Jefferson City, Missouri
  - Western Regional Center for Brain & Spine Surgery, Surgery Center of S. Nevada, Las Vegas, Nevada
  - Buffalo Spine Surgery, Kenmore Mercy, Lockport, New York
  - Duke University Medical Center, Chapel Hill, North Carolina

REFERENCES:
- See also: NuVasive, Inc. — http://www.nuvasive.com